CLINICAL TRIAL: NCT05929963
Title: Observational Study of the Interaction Between Hepatitis C Virus Infection and Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Head of Department, Beijing Ditan Hospital
Other Study IDs: DTXY28
Record Dates: First submitted 2023-05-08; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Hepacivirus; Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HCV Ab(+）HCVRNA（-）: HCV Ab（+） HCVRNA(-) in pregnant women
  Interventions: Other: HCV infection status
- HCV Ab(+）HCVRNA（+）: HCV Ab(+）HCVRNA（+）in pregnant women
  Interventions: Other: HCV infection status
- HCVAb(-) HCVRNA(-): HCV Ab(-）HCVRNA（-）in pregnant women
  Interventions: Other: HCV infection status

INTERVENTIONS:
Other: HCV infection status — Divided into 3 groups based on HCVAb and HCVRNA status

SUMMARY:
The goal of this observational study is to learn about he effects of hepatitis C virus on pregnancy. The main question[s] it aims to answer are:

Effect of hepatitis C virus on liver function in pregnant women Mother-to-child transmission rate in pregnant women with hepatitis C

DETAILED DESCRIPTION:
This study aims to collect demographic data, biochemical indicators during pregnancy, pregnancy complications, and fetal outcomes through the hospital HIS and LIS systems to investigate the impact of HCV infection on pregnancy outcomes, mother-to-child transmission, and long-term child development, and to provide assistance in the clinical management of pregnant women with HCV infection.

ELIGIBILITY:
Inclusion Criteria:

* normal (anti-HCV negative) or RNA negative (anti-HCV positive and HCV RNA negative) or RNA positive (anti-HCV positive and HCV RNA positive) pregnant women
* pregnant women aged 20-45 years
* complete pregnancy data available

Exclusion Criteria:

* Combination of other liver diseases such as viral hepatitis (hepatitis A, B, D, E), alcoholic hepatitis, autoimmune hepatitis, metabolic hepatitis, non-alcoholic fatty liver disease
* Combination of other viral infections with potential loss of liver function
* Mental illness
* Patients with immunosuppression
* Mother with cirrhosis or liver tumour

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women with hepatitis C:RNA negative (anti-HCV positive and HCV RNA negative) or RNA positive (anti-HCV positive and HCV RNA positive) pregnant women
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of various adverse pregnancy outcomes | 2023-2025
  The probability of postpartum haemorrhage, gestational diabetes mellitus and gestational hypertension in pregnant women infected with hepatitis C virus and the associated factors affecting them

SECONDARY OUTCOMES:
Mother-to-child transmission rate of HCV | 2023-2025
  Mother-to-child transmission rate of HCV in pregnant women and correlation with HCV RNA viral load
Development of children born to HCV pregnant women | 2023-2025
  We will follow up on the child's weight (weight in kilograms）, heigh（height in meters）,Body mass index（BMI described in kg/m^2) ,head circumference（Head circumference described in metres），Head up, roll over, sit, crawl, stand and talk start time（Describe time in months）.

CONTACTS AND LOCATIONS:
Overall Officials: Yao Xie, Doctor, Principal Investigator — Beijing Ditan Hospital
Locations (1):
- Beijing Ditan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No